CLINICAL TRIAL: NCT05770167
Title: Effects of Dapagliflozin on Exercise Capacity, Respiratory Function, Biomarkers, Sleep Apnoeas and Left Ventricular Remodelling in Heart Failure Patients
Brief Title: Effects of Dapagliflozin on Cardiorespiratory Parameters in Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1756
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Left Ventricle Remodeling; Sleep Apnea; Cardiopulmonary Exercise Test
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dapagliflozin is a molecule belonging to the class of sodium-glucose transporter type 2 (SGLT2-i) inhibitors. This type of drug, initially used in the treatment of diabetes mellitus, has in recent years demonstrated significant prognostic benefit in patients with heart failure even in the absence of diabetes mellitus. The new international heart failure guidelines have taken up this evidence by suggesting the use of SGLT2-i therapy in patients with heart failure with reduced ejection fraction (HFrEF). Given the drug's recent introduction into clinical routine, the evaluation of "field" experience is important to refine the clinical management of patients treated with SGLT2-i. Moreover, SGLT2-i has currently been shown to be effective in some small preliminary studies in improving ejection fraction and some echocardiographic parameters of ventricular remodelling on top of concomitant optimal medical therapy, although further data are needed in this regard. In particular, the potential benefit of SGLT2-i therapy on exercise capacity, respiratory function parameters, biomarkers and left ventricular remodelling in patients with heart failure has not been extensively studied at present. In this regard, the cardiopulmonary exercise test (CPET) allows the derivation of prognostic functional parameters in patients with chronic heart failure such as peak VO2 and the ventilation/CO2 slope. CPET is a valid, recognised and accurate tool for risk stratification in patients with heart failure. In addition, there are no data available on the effect of SGLT2-i on lung diffusion (DLCO) and specific markers of the alveolar-capillary membrane, such as surfactant binding proteins, as well as on the presence of sleep apnoea, a particularly relevant parameter for the prognosis of decompensated patients.

The aim of the study is to evaluate changes in exercise capacity, spirometry, DLCO, echocardiographic parameters of left ventricular systolic-diastolic function, Nt-proBNP dosage, ST-2, surfactant binding proteins, sleep apnoea, impedance measurement and quality of life in a single-centre cohort of 70 patients with heart failure with stable reduced left ventricular ejection fraction (functional class NYHA II and III) and guideline candidates for treatment with Dapagliflozin.

Patients will undergo, as per regular clinical practice, an initial assessment (baseline) that will include a clinical evaluation, KCCQ questionnaire for quality of life assessment, spirometry, DLCO, impedance measurement, polysomnography, a cardiopulmonary ramp test, blood tests with dosage of Nt-proBNP, ST-2 and surfactant binding protein, and a standard transthoracic echocardiogram. At baseline, the patient will start treatment with Dapagliflozin at the standard dosage of 10mg/day. A similar evaluation with the same study procedures will be performed 6 months after the start of therapy. A re-evaluation of the patient including venous blood sampling is planned between 2 and 4 weeks after the start of Dapagliflozin from clinical practice. In the context of this sampling, the assay of the biomarkers under study will also be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* stable clinical conditions
* Diagnosis of heart failure according to European guidelines (ESC) with EF≤40%
* New York Heart Association Class (NYHA) II-III, despite optimised treatment for heart failure, candidates for treatment with Dapagliflozin according to current guidelines
* Ability to perform cardiopulmonary testing (CPET)
* Patients who have signed written informed consent

Exclusion Criteria:

* Contraindication for Dapaglilozin prescription
* Moderate-severe obstructive pulmonary disease (COPD)
* Estimated glomerular filtrate (eGFR) <30 mL/min/1.73m2 according to MDRD criteria
* Inability or contraindication to perform a CPET
* Taking an investigational drug within 30 days prior to administration of Dapagliflozin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with heart failure with reduced left ventricular ejection fraction, stable (NYHA functional class II and III) and guideline candidates for treatment with Dapagliflozin
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
exercise capacity change | 6 months
  Evaluation of the change in patients' exercise capacity by raising oxygen consumption at peak exercise during cardiopulmonary testing

SECONDARY OUTCOMES:
change in FEV1 | 6 months
  Change in lung function in terms of forced expiratory volume in 1 s FEV1 (spirometry)
change in DLCO | 6 months
  Change in lung function in terms of DLCO (lung diffusion capacity for carbon monoxide)
Change in Nt-proBNP | 6 months
  Change in blood levels of heart failure biomarker Nt-proBNP (amino terminal pro-B-type natriuretic peptide)
Change in ST-2 | 6 months
  Change in blood levels of heart failure biomarker ST-2 (soluble interleukin 1 receptor-like 1)
Change in surfactant binding protein | 6 months
  Change in blood levels of biomarker surfactant binding protein
change in LVEF | 6 months
  Chnage in left ventricular ejection fraction (echocardiography)
change in left ventricular volumes | 6 months
  Change in left ventricular volumes (echocardiography)
change in central sleep apnoeas | 6 months
  Change in central sleep apnoeas (Nocturnal cardiorespiratory monitoring)
change in quality of life | 6 months
  Change in patients' quality of life evaluated through Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
change in hydration index | 6 months
  Change in hydration index HI assessed through Bioimpedance vector analysis (BIVA)
population stratification according to VO2 peak higher and lower than 15 ml/min/kg | 6 months
  Show any differences in clinical response depending on the severity of heart failure (stratified according to VO2 peak higher and lower than 15 ml/min/kg at CPET)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Mapelli, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy